CLINICAL TRIAL: NCT06708169
Title: Effect of Preemptive Education on the Incidence of Maternal Intraoperative Shivering in Elective Cesarean Delivery: a Randomized Controlled Trial
Brief Title: Effect of Preemptive Education on the Incidence of Maternal Intraoperative Shivering in Elective Cesarean Delivery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2408-040-1558
Record Dates: First submitted 2024-10-31; First posted 2024-11-27 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2024-09

CONDITIONS: Shivering; Spinal Anesthesia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patients without preoperative education by anesthesiologists (No Intervention): Patients get minimal information about the surgical process and their questions will be answered by obstetrician.
- Patients with preoperative education by anesthesiologists (Experimental): Patients get preemptive education about the whole process from anesthesia to recovery stage within 15 minute by anesthesiologists.
  Interventions: Behavioral: preemptive education provided by anesthesiologists

INTERVENTIONS:
Behavioral: preemptive education provided by anesthesiologists — A preemptive education about 4 stages (prepare, anethesia, surgery, and recovery) by anesthesiologists within 15 minute.
  Arms: Patients with preoperative education by anesthesiologists

SUMMARY:
The goal of this study is to learn about the effect of preemptive education on reducing intraoperative maternal shivering in elective cesarean delivery. The main question it aims to answer is:

Does preemptive education by anesthesiologists reduce intraoperative maternal shivering in elective cesarean delivery?

ELIGIBILITY:
Inclusion Criteria:

* Age 19 years or older
* Gestational age 37 weeks or above
* Elective surgey

Exclusion Criteria:

* Emergency surgery
* Any sign of onset of labor
* Difficulty with communication
* Contraindications of spinal anesthesia
* Pre-eclampsia

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2024-12-09 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with intraoperative maternal shivering | From the moment the patient enters the operating room (0 minute) until leaving the operating room on the same day, expected to be up to 180 minutes.
  Record when shivering occurred within the time frame

SECONDARY OUTCOMES:
Intraoperative body temperature | 0, 15, 30, 45, 60, 75, 90, 105, 120, 135, 150, 165, 180 minutes after entering the operating room until the end of surgery.
Intraoperative pain (Numeric rating scale, NRS). | From the moment the patient enters the operating room (0 minute) until leaving the operating room on the same day, expected to be up to 180 minutes.
  NRS 0: no pain 1-3: mild pain (nagging, annoying, interfering little with acitivities of daily living (ADLs)) 4-6: moderate Pain (interferes significantly with ADLs) 7-10: severe Pain (disabling; unable to perform ADLs)
  Record when the patient complained pain within the time frame
Spinal anesthesia level (dermatome) | From the intrathecal injection (0 minute) until at the end of surgery (0, 5, 10, 25, 40, 55, 75 minute, at the end of surgery)
Post-operative spinal anesthesia level in recovery room | From the time the patient enters the recovery room (0 minute) until leaving the recovery room (0, 15, 30, 45 minute, at the time the patient leaves the recovery room)
  The level(dermatome) of spinal anesthesia will be checked by pin-prick test by an anesthesiologist or nurse.
Number of Participants with Post-operative shivering in recovery room | From the time the patient enters the recovery room (0 minute) until leaving the recovery room (0, 15, 30, 45 minute, at the time the patient leaves the recovery room)
Post-operative body temperature in recovery room | From the time the patient enters the recovery room (0 minute) until leaving the recovery room (0, 15, 30, 45 minute, at the time the patient leaves the recovery room)
Post-operative nausea and vomiting in recovery room (by questionnaire) | From the time the patient enters the recovery room (0 minute) until leaving the recovery room (0, 15, 30, 45 minute, at the time the patient leaves the recovery room)
  Nausea and vomiting will be assessed by questionnaire. (yes/no)
Patient's satisfaction by questionnaire | From the end of surgery until 24 hours after surgery
  Patient's satisfaction about pre-operative preparation, anesthesia, and surgery by questionnaire.
  Participants will respond their satisfaction by score 0-10. (A higher score means higher satisfaction. )
Pain (assessed by NRS) until post-operative day 1 | At 6, 12, 18, 24 hours after the end of surgery
  NRS (numeric rating scale) is detailed at Outcome number 3.
Analgesic dosage (Morphile miligram equivalents) until post-operative day 1 | From the end of surgery until 24 hours after surgery
Obstetric quality of recovery until post-operative day 1 | At 24 hours after surgery
  Quality of recovery will be assessed by Obstetric Quality of Recovery-11K survery, which is a questionnaire completed by participants.
  Higher score means higher quality of recovery.

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, Jongno-gu, South Korea